CLINICAL TRIAL: NCT02156713
Title: Constraint Induced Movement Therapy Summer Camp for Children With Unilateral Cerebral Palsy Ages 3-7
Brief Title: Constraint Induced Movement Therapy Summer Camp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kelly Tanner (Other)
Responsible Party: Sponsor-Investigator, Kelly Tanner, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB14-00197
Record Dates: First submitted 2014-06-02; First posted 2014-06-05 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Cerebral Palsy; Cerebral Palsy, Diplegic, Infantile
Keywords: Hemiparesis; Occupational Therapy
MeSH Terms: conditions — Cerebral Palsy; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CIMT Camp (Experimental): Members of this study will participate in the group CIMT camp.
  Interventions: Behavioral: CIMT Camp

INTERVENTIONS:
Behavioral: CIMT Camp

SUMMARY:
Constraint induced movement therapy (CIMT) is an intervention for unilateral cerebral palsy (CP). It is currently part of standard of care for children with unilateral CP, but is typically done one-on-one and with the child wearing a cast 24 hours a day during the duration of treatment. The purpose of this study is to assess the effects of an intensive group-based CIMT summer camp in which participants wear a removable cast on upper extremity function, occupational performance, and patient-specific goals. The investigators hypothesize that upper extremity skills and occupational performance will increase, and that patients will reach their individualized goals.

ELIGIBILITY:
Inclusion Criteria:

* Scores of level I, II or III on the Manual Ability Classification System
* Independent grasp
* Ability to ambulate independently or with an assistive device
* Sufficient cooperation and cognitive understanding to participate in a group.

Exclusion Criteria:

* Lack of hand function
* Fixed contractures
* Active seizures
* High tone
* Medical instability
* Non-English speaking parents.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in Canadian Occupational Performance Measure Score | Week 5
  The Canadian Occupational Performance Measure asks parents to rate their child's level of occupational performance as well as how satisfied they are with it both before and after treatment.
Goal Attainment Scaling | Week 5
  Parents and therapists identify appropriate goals for the child to achieve at the end of therapy. The therapist then identifies "levels of attainment" for each individual goal.
Change in Manual Ability Classification System Level | Week 5
  The Manual Ability Classification System is an observation-based measure of upper extremity function in individuals with cerebral palsy.
Change in Pediatric Motor Activity Log Score | Week 5
  This caregiver questionnaire addresses how often and how well a child uses his or her affected extremity outside of the therapy setting.
Change in Quality of Upper Extremity Skills Test Score | Week 5
  This is an observation-based measure during which the therapist evaluates the quality of an individual's upper extremity movement with regard to dissociated movement, grasp, protective extension, and weight bearing.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly J Tanner, MOT, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States